CLINICAL TRIAL: NCT00506311
Title: A Randomized Trial Evaluating the Use of Fibrin Tissue Adhesive Following Superficial Groin Dissection in Patients With Melanoma
Brief Title: Evaluating the Use of Fibrin Tissue Adhesive in Melanoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS01-564
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Melanoma
Keywords: Superficial Groin Dissection; Melanoma; Fibrin Tissue Adhesive; Fibrin Sealant; Tisseel; Seroma
MeSH Terms: conditions — Melanoma; Seroma | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fibrin Sealant (Experimental)
  Interventions: Drug: Fibrin Sealant
- No Fibrin Sealant (No Intervention)

INTERVENTIONS:
Drug: Fibrin Sealant — Tisseel applied externally to the dissected groin area.
  Other Names: Tisseel
  Arms: Fibrin Sealant

SUMMARY:
Primary Objective:

1. To determine whether the use of a fibrin sealant applied to superficial groin soft tissues following node dissection can result in decreased cumulative postoperative drainage, earlier drain removal, and lower incidence of seroma.

Secondary Objectives:

1. To determine the postoperative morbidity rate using fibrin sealant following superficial groin dissection.
2. To assess patient-valuation of outcome by performing a cost-benefit analysis using a willingness-to-pay model.
3. To determine if serum levels, lymphatic fluids level, or cutaneous expression of vascular endothelial growth factor-D (VEGF-D), vascular endothelial growth factor-C (VEGF-C) or their receptor, vascular endothelial growth factor receptor-3 (VEGFR-3) correlates with nodal tumor burden or development of lymphedema in patients with melanoma.

DETAILED DESCRIPTION:
Patients in this study are scheduled to have groin dissection as part of their surgery for treatment of their melanoma.

Within 2 weeks before entry into the study, patients will have a complete physical exam and medical history.

These patients will be randomly assigned (as in the toss of a coin) to one of two groups. Patients in one group will receive TISSEEL applied externally to the dissected groin area. Patients in the other group will receive no fibrin sealant.

For patients who are admitted to the hospital, the surgical site will be monitored by the surgeon for evidence of wound complications in the first 24 hours after surgery. At the time of discharge from the hospital, patients will be instructed in drain care and how to measure the drainage each day until the drain is removed.

The contents of the drain will be collected from patients during the first day after surgery, during the first return follow-up visit to M.D. Anderson Cancer Center, and during drain removal.

Follow-up wound exams will be performed by the local primary physician or in the M.D. Anderson Melanoma Clinic between 1-4 weeks and 6 weeks after surgery. Participation will be over after the 6-week follow-up.

This is an investigational study. The sealant is FDA approved, though its use in this study is experimental. About 58 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Part I - Inclusion Criteria Patients that consent to participate.
* Patients with melanoma who have undergone superficial node dissection (with or without a concurrent deep (ilioinguinal) node dissection within the last six months as part of their surgical treatment will be considered for the study.
* Part II- Inclusion Criteria Patients that consent to participate.
* Patients with melanoma for which a superficial node dissection is indicated (with or without a concurrent deep (ilioinguinal) node dissection.

Exclusion Criteria:

* Part II - Exclusion Criteria Patients with known hypersensitivity to bovine proteins.
* Patient has undergone prior radiation therapy to the operative site (groin).
* Patient is pregnant or lactating.
* Patient is steroid dependent within last 6 months.
* Patient has used aspirin or other anti-platelet drug (excluding Celebrex) within seven days of operation.
* Patients with pre-existing lymphedema.
* Patients with other pre-existing medical conditions as per the discretion of the principal investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2003-02; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Time-to-Drain Removal | From surgery to 30 days post surgery
  The superficial groin drain will be removed once cumulative serous drainage volume 30 ml / 24 hours for 2 days or maximum of = or < 30 days has elapsed since surgery. Time calculated as days from installation of drain at first day of surgery to removal.

CONTACTS AND LOCATIONS:
Overall Officials: Janice N. Cormier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Mortenson MM, Xing Y, Weaver S, Lee JE, Gershenwald JE, Lucci A, Mansfield PF, Ross MI, Cormier JN. Fibrin sealant does not decrease seroma output or time to drain removal following inguino-femoral lymph node dissection in melanoma patients: a randomized controlled trial (NCT00506311). World J Surg Oncol. 2008 Jun 18;6:63. doi: 10.1186/1477-7819-6-63. PMID 18564433
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org